CLINICAL TRIAL: NCT02709616
Title: Personalized Cellular Vaccine Therapy in Treating Patients With Newly Diagnosed Glioblastoma (PerCellVac)
Brief Title: Personalized Cellular Vaccine for Glioblastoma (PERCELLVAC)
Acronym: PERCELLVAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong 999 Brain Hospital (Other)
Collaborators: Jinan University Guangzhou (Other); Beijing Tricision Biotherapeutics Inc (Industry); Zhuhai Trinomab Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jian Zhang, Jian Zhang, MD, Professor, Vice President of Guangdong 999 Brain Hospital, Chairman, Department of Surgery, Guangdong 999 Brain Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ag-mRNA-DC-999brain
Record Dates: First submitted 2016-03-07; First posted 2016-03-16 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; DC vaccine; tumor antigen; personalized vaccine
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Personalized cellular vaccine (Experimental): DC based cellular vaccine
  Interventions: Biological: Personalized cellular vaccine

INTERVENTIONS:
Biological: Personalized cellular vaccine — Biological: DC-based cellular vaccine. Subjects will undergo surgical resection and standard 6-week chemo/radiotherapy and cycles of TMZ treatment. They will receive biweekly cellular vaccines.
  Other Names: Tumor antigen pulsed DC vaccine

SUMMARY:
Dendritic cell-based cellular vaccine for tumor therapy has shown efficacy. This study is designed to perform a personalized clinical trial by first analyzing the expression of tumor associated antigens in patients with newly diagnosed glioblastoma and then immunizing the patients with personalized DC-based cellular vaccine. Immune responses to tumor antigens will be monitored. Safety and efficacy will be observed in the study.

DETAILED DESCRIPTION:
This is an open label, single-arm, single-institution, Phase I study designed to investigate the safety and efficacy of personalized cellular tumor vaccine for patients with newly diagnosed glioblastoma (GBM). Newly diagnosed GBM patients will undergo tumor resection. The tumors will be analyzed for the expression of a panel of glioma-associated antigens and immune-related genes. Post surgical treatment will be 6 weeks standard chemotherapy with temozolomide and concurrent radiotherapy and continue cycles of temozolomide within a 28-day window. Patients will undergo leukapheresis either after surgery or after concurrent radio/chemotherapy. Based on individual tumor antigen expression, in vitro transcribed mRNA will be generated and used to pulse in vitro generated DCs. The patients will be immunized i.d. and i.v. biweekly with DC cellular vaccines. Safety and efficacy will be monitored. The primary objective is to assess the safety of the personalized cellular vaccines. The secondary objective is to assess the specific T cell response to immunized vaccines. In addition, the antitumor efficacy of the vaccines will be measured using iRANO criteria, progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed glioblastoma grade IV
* Patients at the age of 18-65.
* Patients must have undergone maximal surgical resection of the tumor.
* Patients with Karnofsky scores > or =70
* Patients with normal range of hematologic and metabolic test results.
* Patients must have no corticosteroids treatment at least one week before vaccination.
* Patients capable of understanding the study and signed informed consent.

Exclusion Criteria:

* Breast feeding females.
* Pregnant women.
* Infectious diseases HIV, HBV, HCV
* Documented immunodeficiency
* Documented autoimmune disease
* Any serious or uncontrolled medical or psychiatric conditions, for example, severe pulmonary, cardiac or other systemic disease.
* Patient inability to participate as determined by PI discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events and severe adverse events [safety and Tolerability] | 3 years since the beginning of the first vaccine
  Incidence of adverse events and severe adverse events to measure safety and tolerability of mRNA-TAA pulsed autologous DC cellular vaccine

SECONDARY OUTCOMES:
Antitumor antigen specific T cell response | 4 weeks after the last vaccine
  The frequency of peripheral CD8+ and CD4+ T cell response to the vaccine.
Progression-free survival | 12 months since the beginning of the first vaccine.
  Progression-free survival will be monitored for 1year.
Overall survival | 3 years since the beginning of the first vaccine
  Overall survival will be monitored for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, M.D., Principal Investigator — Guangdong 999 Brain Hospital
Locations (1):
- Guangdong 999 Brain Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wang QT, Nie Y, Sun SN, Lin T, Han RJ, Jiang J, Li Z, Li JQ, Xiao YP, Fan YY, Yuan XH, Zhang H, Zhao BB, Zeng M, Li SY, Liao HX, Zhang J, He YW. Tumor-associated antigen-based personalized dendritic cell vaccine in solid tumor patients. Cancer Immunol Immunother. 2020 Jul;69(7):1375-1387. doi: 10.1007/s00262-020-02496-w. Epub 2020 Feb 20. PMID 32078016
- See also: Publication of the trial results — https://pubmed.ncbi.nlm.nih.gov/32078016/